CLINICAL TRIAL: NCT02989493
Title: Randomized Controlled Trial Targeting Noradrenergic Stress Mechanisms in Alcoholism With Doxazosin
Brief Title: Testing Doxazosin to Treat Stress Mechanisms in Alcoholism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015-1009; R01AA024388 (NIH); A487400 (Other: UW Madison); L&S\PSYCHOLOGY\PSYCHOLOGY (Other: UW Madison); Protocol Version 11/7/2019 (Other: UW Madison)
Record Dates: First submitted 2016-12-01; First posted 2016-12-12 (Estimated); Results first posted 2021-03-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Alcoholism
Keywords: Alcoholism; Stress; Norepinephrine; Doxazosin; Anxiety; Startle Potentiation; Relapse; Adrenergic Antagonists; Surrogate Endpoint
MeSH Terms: conditions — Alcoholism; Anxiety Disorders; Recurrence | interventions — Doxazosin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Doxazosin (Experimental): Participants receive 8 weeks of doxazosin (8mg target dose).
  Interventions: Drug: Doxazosin
- Placebo (Placebo Comparator): Participants will receive 8 weeks of matched placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Doxazosin — Doxazosin
  Arms: Doxazosin
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Double-blind, placebo controlled, randomized controlled trial (RCT) for Alcohol Use Disorder examining the effects of doxazosin, a norepinephrine alpha1 receptor antagonist, on stress reactivity and clinical outcomes.

DETAILED DESCRIPTION:
OBJECTIVES:

1. To translate the preclinical evidence from animal models to stress-induced relapse in humans via direct pharmacological antagonism of the noradrenergic system in abstinent alcoholics with doxazosin, an alpha1 noradrenergic receptor blocker.
2. To screen the efficacy of doxazosin to target stress-related relapse mechanisms in abstinent alcoholics as a cost-effective first step to repurpose this alpha1 noradrenergic antagonist for relapse prevention in addiction.

PARTICIPANTS:

136 participants with an Alcohol Use Disorder in early abstinence.

STUDY OVERVIEW:

136 adults with an Alcohol Use Disorder in early abstinence (1-8 weeks abstinent) will participate in a randomized controlled trial (RCT) to examine the efficacy of 8 mg doxazosin (vs. placebo, between-subjects) on stress reactivity and clinical outcome measures (e.g., drinks/week, alcohol craving) during a 8 week treatment period. Doxazosin's impact on stress-related relapse mechanisms will be assessed using a well-validated human model of stressor reactivity (No Shock, Predictable Shock, Unpredictable Shock [NPU] task) at baseline (pre-treatment) and after 4 weeks of treatment. The NPU task has strong translational ties to both methods (e.g., unpredictable vs. predictable electric shock) and measures (e.g., startle potentiation) from the preclinical literature in animals. This laboratory stress task serves as an attractive early surrogate endpoint post-treatment to assess treatment efficacy and examine stress mechanisms.

AIMS and HYPOTHESIS:

AIM 1: Examine effects of a therapeutic dose of doxazosin on responses to unpredictable stressors in NPU task. The aim is to obtain preliminary evidence via a laboratory surrogate endpoint to repurpose doxazosin for the treatment of stress-induced relapse mechanisms in alcoholism.

PREDICTIONS: Following four weeks of therapeutic dosing, doxazosin (8 mg vs. placebo, between-subjects) will selectively reduce response to unpredictable (vs. predictable) stressors indexed by physiological defensive reactivity (startle potentiation) and self-reported negative affect and craving in abstinent alcoholics.

AIM 2: Examine effects of a therapeutic dose of doxazosin on early clinical outcome measures. The aim is to obtain additional evidence via clinical outcome measures to repurpose doxazosin for the treatment of stress-induced relapse mechanisms in alcoholism.

PREDICTIONS: Following eight weeks of therapeutic dosing, doxazosin (8 mg vs. placebo, between-subjects) will increase continuous abstinence and decrease drinking days per week and drinks per week during the medication treatment period. Doxazosin will also decrease craving measured during the 8th week of medication use when participants have achieved the maximum dose for 4.5 weeks.

AIM 3: Examine predictive validity of pre-treatment laboratory tests of noradrenergic relevant stress-reactivity on surrogate endpoint and clinical outcome measures. The aim is to link individual differences in stress reactivity at baseline (i.e. pre-treatment) to laboratory surrogate endpoints and early clinical outcome measures following therapeutic dosing.

PREDICTIONS: Higher pre-treatment reactivity during unpredictable stressors will predict poorer surrogate endpoint and clinical outcomes overall. Therapeutic 8 mg dose effects of doxazosin will be greater among alcoholics who display higher pre-treatment reactivity to unpredictable stressors.

AIM 4: Examine if the effects of doxazosin on clinical outcome measures are mediated by a reduction of stress-reactivity as measured by the NPU task. The aim is to identify whether reductions in stress-reactivity (NPU task) is the mechanism through which doxazosin has its effect on drinking behavior (clinical outcome).

PREDICTIONS: The direct effect of doxazosin (vs. placebo) following 8 weeks of therapeutic 8 mg dosing on clinical outcomes (e.g., continuous abstinence, drinking days/week, drinks/week) will be partially mediated by the indirect effect of doxazosin on surrogate endpoint of NPU stress reactivity at 4 weeks.

ELIGIBILITY:
INCLUSION CRITERIA:

* Diagnostic and Statistical Manual (DSM-5) diagnosis of Alcohol Use Disorder, Moderate-Severe
* Alcohol abstinent for 1 - 8 weeks
* Ages of 18 to 65

Exclusion criteria are divided into three broad categories of Medical, Psychiatric/Behavioral, and Medications/Therapies.

EXCLUSION CRITERIA: Medical

* Blood alcohol concentration above 0.00.
* Color blind.
* Heart rate >100 beats per minute after five minutes seated.
* Heart rate <55 beats per minute after five minutes seated.
* Systolic BP <100 after five minutes seated.
* Systolic BP drop >20mm Hg or diastolic BP drop >10mm Hg after two minutes standing.
* Dizziness, lightheadedness, unsteadiness or other problems (e.g, nausea, blurry vision) after two minutes standing.
* Uncorrected auditory/vision problems.
* Current treatment for chronic pain condition.
* Past or current coronary artery disease, cerebrovascular accident, congestive heart failure.
* Current chronic renal insufficiency, liver insufficiency or moderate hepatic impairment, pancreatitis, immunosuppressive therapy, or cancer with systemic effects or therapy.
* Benign positional vertigo, Meniere's disease, or narcolepsy.
* Previous allergic or adverse reaction to doxazosin or other alpha1 noradrenergic antagonist.
* Scheduled or reported plans for cataract surgery prior to study completion.
* Currently symptomatic of alcohol withdrawal [Clinical Institute Withdrawal Assessment for Alcohol, revised (CIWA-Ar) Score > 10, or positive for any 'visual, auditory or tactile disturbances,' or for 'orientation and clouding of sensorium']
* Discharged from inpatient treatment for Alcohol Use Disorder or alcohol detoxification within past 7 days.
* Currently medically unstable.
* Electrocardiogram (ECG) clinical over-read indicates concerns of cardiac function.
* Other self-reported acute or unstable illness that, in the opinion of the study team, would preclude a safe and reliable study participation

EXCLUSION CRITERIA: Female Participants Only

* Non-negative urine pregnancy test.
* Women of childbearing potential (see definition below) must agree to use one of the following forms of birth control until after study completion. Acceptable birth control is defined as the following methods of contraception: abstinence; hormonal contraceptives (e.g. combined oral contraceptives, patch, vaginal ring, injectables, and implants); intrauterine device (IUD) or intrauterine system (IUS); vasectomy of partner and tubal ligation; "single" barrier methods of contraception (e.g. male condom, female condom, cervical cap, diaphragm, contraceptive sponge) with use of spermicide; or "double barrier" method of contraception (e.g. male condom with diaphragm, male condom with cervical cap).
* Breastfeeding.

NOTE: Women of childbearing potential are females who have experienced menarche and do not meet the criteria for women not of childbearing potential. Women not of childbearing potential are females who are permanently sterile (e.g., hysterectomy, bilateral oophorectomy) or postmenopausal. Postmenopausal is defined as 12 consecutive months with no menses without an alternative medical cause.

EXCLUSION CRITERIA: Psychological/Behavioral

* Self-reported lifetime diagnosis of schizophrenia, schizoaffective disorder, psychotic disorder not otherwise specified, bipolar disorder (with manic episode), borderline personality disorder, or any neurocognitive disorder that may impair a reliable, safe participation.
* Current suicidal ideation.
* Current active substance use disorder other than alcohol or tobacco.

EXCLUSION CRITERIA: Medications/Therapies

* Currently prescribed or used within past week: doxazosin or other alpha1 noradrenergic antagonist (e.g., prazosin, terazosin).
* Currently prescribed or used within past week: substances with stimulant properties (e.g., d-amphetamine, methylphenidate, ephedra, pseudoephedrine).
* Currently prescribed or used within past week: Sildenafil (Viagra), tadalafil (Cialis), and vardenafil (Levitra).
* Currently prescribed or used within past week: beta-blockers (e.g., propanolol), alpha2 agonists (e.g., clonidine, guanfacine, dexmedetomidine), and serotonin and norepinephrine reuptake inhibitors (SNRI) (e.g., venlafaxine, duloxetine, atomoxetine, viloxazine).
* Currently used daily or used within past week: alpha1 agonists (e.g., midodrine, metaraminol, oxymetazoline, phenylephrine).
* Currently used daily or used within past week: Benzodiazepines (e.g., diazepam, chlordiazepoxide, lorazepam, clonazepam, alprazolam), zolpidem (Ambien), zaleplon (Sonata), zopiclone (Imovane), eszopiclone (Lunesta), doxepin (Silenor).
* Currently prescribed and used daily or used within past 2 weeks: Trazodone.
* Currently prescribed or used within 2 weeks: Disulfiram (Antabuse).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John J Curtin, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available online upon study completion at the Open Science Framework: https://osf.io

REFERENCES:
- See also: Dr. John Curtin's Addiction Research Center — http://arc.psych.wisc.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled via community advertisement and clinical referral.
Pre-assignment Details: 61 participants were consented, passed medical screening, and were assigned to a drug group.
Period: Overall Study
Arm/Group | Doxazosin | Placebo
Started | 29 | 32
Completed | 29 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Doxazosin | Placebo | Total
Number analyzed (Participants) | 29 | 32 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] — self report age
  years | 45.6 (11.9) | 39.7 (10.8) | 42.5 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 23 | 23 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 28 | 30 | 58
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 27 | 27 | 54
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — All participants were enrolled in Madison, WI, USA
  participants
    United States | 29 | 32 | 61

OUTCOME MEASURES:

1. Primary Outcome: Startle Potentiation During Stress Reactivity Task
Description: Startle potentiation is used to study anxiety and fear with No-shock, Predictable-shock, Unpredictable-shock (NPU) task; a common, well-validated laboratory stressor task. In the Predictable condition of the NPU task, shocks are 100 percent predictable and occur at a consistent, known time. In the Unpredictable condition of the NPU task, shocks are fully unpredictable. A higher score on startle potentiation means a higher stress reactivity response for the given condition.
Time Frame: 4 weeks
Population: Although all 61 participants were able to provide TLFB data through the end of 8 weeks, the NPU task required that they attend a study visit at 4 weeks. 24 participants (10 in doxazosin, 13 in placebo) did not complete that study visit and so have data missing for this outcome measure. 1 (doxazosin) attended the visit but chose not to complete the NPU task. 2 participants (both placebo) completed NPU at this visit, but their NPU data was unusable for this analysis due to technical issues.
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | Doxazosin | Placebo
Number analyzed (Participants) | 18 | 17
microvolts
  Unpredictable startle potentiation | 22.25 (20.18) | 20.76 (23.21)
  Predictable startle potentiation | 26.22 (30.90) | 22.21 (35.93)

2. Primary Outcome: Number of Participants Reporting Any Heavy Drinking Days
Description: Timeline-followback (TLFB) was administered twice at 4 weeks and 8 weeks. Participants reported the number of drinks per day for each previous 30 day period. Any heavy drinking was scored "yes" if participant reported any days of heavy drinking (> 4/3 standard drinks for men/women) during the total 8 week assessment period; "no" if no heavy drinking was reported
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Doxazosin | Placebo
Number analyzed (Participants) | 29 | 32
Participants | 17 | 21

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Doxazosin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/32
Other Adverse Events (participants affected / at risk) | 24/29 | 28/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Doxazosin (N=29) | Placebo (N=32)
Orthostatic hypertension (Vascular disorders) | 14 (24) | 7 (18)
Dizziness (Ear and labyrinth disorders) | 9 (17) | 7 (9)
Cardiac arrhythmia (Cardiac disorders) | 8 (12) | 6 (7)
Chest pains (Cardiac disorders) | 2 (5) | 0 (0)
Fatigue (General disorders) | 15 (38) | 17 (36)
Edema (Cardiac disorders) | 3 (6) | 0 (0)
Rhinitis (General disorders) | 13 (29) | 5 (9)
Headache (General disorders) | 9 (25) | 11 (17)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (5)
Dry mouth (General disorders) | 10 (30) | 8 (15)
Nausea or diarrhea (Gastrointestinal disorders) | 9 (14) | 8 (9)
Blurry vision (Eye disorders) | 4 (4) | 0 (0)
Polyurea (Renal and urinary disorders) | 2 (6) | 4 (8)
General symptoms, nonspecific (General disorders) | 8 (9) | 6 (10)
Priapism (Reproductive system and breast disorders) | 2/19 (2) | 0/20 (0) — This was only assessed in men

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-07): https://cdn.clinicaltrials.gov/large-docs/93/NCT02989493/Prot_SAP_000.pdf